CLINICAL TRIAL: NCT03714074
Title: Patient Satisfaction, Peri-implant Parameters and Crestal Bone Evaluation of PEEK (Polyetheretherketone) Abutments Versus Zirconium Abutments Restored With PEEK Based Superstructure: A Randomized Clinical Trial
Brief Title: Patient Satisfaction, Peri-implant Parameters and Crestal Bone Evaluation of PEEK (Polyetheretherketone) Abutments Versus Zirconium Abutments Restored With PEEK Based Superstructure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Ali youssef, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-09-27
Record Dates: First submitted 2018-09-25; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Patients Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEK abutment (Experimental): PEEK abutment restored with PEEK superstructure
  Interventions: Device: PEEK implant abutment
- Zirconia abutment (Experimental): zirconia abutment restored with PEEK superstructure
  Interventions: Device: Zirconia abutment

INTERVENTIONS:
Device: PEEK implant abutment — Implants will be restored with abutments made from polyetheretherketone (PEEK) abutments and a PEEK superstructure
  Other Names: Polyetheretherketone abutments
  Arms: PEEK abutment
Device: Zirconia abutment — Imolants will be restored with zirconia abutments and a PEEK superstructure
  Other Names: esthetic abutment, hybrid abutment, all ceramic abutment
  Arms: Zirconia abutment

SUMMARY:
The aim of the study is to evaluate the patients' satisfaction, peri-implant parameters (bleeding on probing, probing depth and plaque index) and crestal bone resorption of implants restored with PEEK abutments restored with PEEK superstructure compared to implants restored with zirconia abutments with PEEK superstructure.the NULL HYPOTHESIS;There is no difference between the two groups

DETAILED DESCRIPTION:
Trial design:

Randomized Controlled Trial., Parallel Design., Allocation ratio 1:1

This study will be carried out on patients enrolled from the Outpatient clinic in the Fixed Prosthodontics clinic, Faculty of Dentistry, Cairo University.

First Visit: ( Diagnosis and records Making)

Patients will be recalled to the outpatient clinic, treatment will be discussed with the patient in details with the expected timeline and full duration of the treatment and a signed consent will be obtained from the patient.

Thorough medical history will be taken from the patient to identify any causes preventing the patient from undergoing the surgery and to eliminate any risk factors. Primary alginate impressions and bite registration will be made to obtain mounted study casts for case study, intra-oral photographs will be taken and the patient will be asked for a CBCT for the area of interest to be studied and discussed .

Second visit: (Implant insertion)

The patient will be locally anaesthetized using Articaine 4% (Septanest, France) , and patient will be left for 5 -10 minutes after which he/she will be examined for objective/subjective signs. If the patient shows any signs of pain or discomfort during examination, another carpule will be administrated.

A full thickness flap will be opened at the surgical site using #15 blade with a sub-crestal incision to expose the crest of the bone and two vertical releasing incisions. The flap will be reflected using a mucoperiosteal elevator. Sequential drilling will be performed according to the desired implant diameter using the drills provided by the surgical kit and the implant will be inserted manually into the osteotomy using the ratchet wrench and driver. The initial stability of the implant will be tested with the torque wrench and the implant opening will be closed using a cover screw. A peri-apical radiograph will be taken to confirm the implant position and assure it is away from vital structures by 2mm.

Flap will be repositioned using a tissue forceps and suturing will be done to secure the flap in position using a 4-0 silk suture material.

Patient will be given the post-operative instructions and hygiene measures and Augmentin 1gm / 12 hours for 7 days and analgesics ( Brufen 400 mg when needed)

Third visit: (Re-entry)

After three to four months, the patient will be recalled for the 2nd stage surgery and implant exposure. Peri-apical radiographs and intra-oral photographs will be taken. The patient will be anaesthetized and the implant will be exposed by a crestal incision using a #15 blade. The cover screw will be replaced with a healing collar which will be left for 2 weeks.

Fourth visit: (Impression making):

After 2 weeks the healing collar will be removed and the transfer copings will be placed for impression making, after setting the impression will be disinfected and send to the laboratory along with the implant replicas for fabrication of the abutments and the prosthesis. The healing collar is replaced till the next visit.

Fifth visit: ( Delivery of the final restoration)

The healing collar will be removed and the abutment and final restoration will be placed over the implant, a peri-apical radiographs will be taken to ensure tightening of the abutment screw and absence of any gaps. Patient will be given oral hygiene instructions

Relevant care/interventions that will be permitted or prohibited during the trial:

* Patients will receive antibiotics and pain killers after the implant insertion
* Patients will be educated with proper hygiene measures and motivated to keep good oral hygiene
* Patients will be advised to stop/ decrease the frequency of smoking to maximum one pack per day and will be prohibited from drinking alcohol.

Primary outcome:

Patients' satisfaction will be measured used the Visual analogue scale; a numerical scale from 0-10 with 0 being the lowest value (dis-satisfied) and 10 being the highest (highly satisfied). The patient will be asked to fill the VAS at time of crown delivery (0) , 3months, 6 months and 12 months

Secondary outcome: will be assessed at 0,3,6 and 12 months

1. Bleeding on Probing Visual Inspection combined with Plastic Periodontal Probe 2 Binary (Yes or No)
2. Probing Depth Graduated periodontal probe 2 Millimeters (m.m)
3. Plaque accumulation Visually 2 Binary (Yes & No)

Tertiary outcome:

Will be assessed at 0,3,6 and 12 months using the standardized peri-apical radiographs and image super-imposition on the software to measure the difference in bony crest height.

Where 0= time of prosthesis delievery.

ELIGIBILITY:
Inclusion Criteria:

1. patients above 18 years old
2. Patients able to read and sign the informed consent.
3. Medically free patients or with controlled systemic condition.
4. Missing tooth/teeth in the esthetic zone
5. Minimum bucco-lingual bone width of 6mm, evaluated using CBCT.
6. Good oral hygiene and favourable occlusion
7. Cooperative and motivated Patients.

Exclusion Criteria:

1. Under 18 years old
2. Illiterate, unable of comprehending or signing the informed consent form
3. Uncontrolled systemic disease (e.g. Diabetes or hypertension) or debilitated health condition
4. Pregnancy
5. Poor oral hygiene or unfavorable occlusion
6. Uncooperative, not willing to return for follow up visits
7. Insufficient bone quantity or quality for implant placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
change in Patients satisfaction: VAS | baseline, 3, 6 and 12 months (1 year)
  Visual analogue scale (VAS) a numerical scale from 0 - 10 , 0 = not satisfied and 10 = highly satisfied

SECONDARY OUTCOMES:
Change in bleeding in probing | baseline, 3 , 6 and 12 months (1 year)
  inserting periodontal probe in gingival sulcus to detect bleeding (yes or no)depth (millimeters)
Change in periodontal probing depth | baseline, 3 , 6 and 12 months (1 year)
  inserting a graduated periodontal probe to detect presence or absence of pockets (yes or No)
Change in Plaque accumilation | baseline, 3 , 6 and 12 months (1 year)
  visual inspection for plaque accumilation (yes or No)

OTHER OUTCOMES:
change in crestal bone resorption | baseline, 3 , 6 and 12 months (1 year)
  in millimeters by superimposition of standerdized radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Amina Zaki, Professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided